CLINICAL TRIAL: NCT04267289
Title: Happy@Home: Delivering Internet-based Cognitive Behavioral Therapy With Homecare Workers to At-Home Seniors
Brief Title: Happy@Home: Delivering iCBT With Homecare Workers to At-Home Seniors
Acronym: Happy@Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Xiaoling Xiang, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2748II
Record Dates: First submitted 2020-02-07; First posted 2020-02-12 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iCBT treatment group (Experimental): Subjects were given license to use Beating the Blues, a commercially available iCBT program. Subjects were given 3 months to use the program.
  Interventions: Behavioral: Beating the Blues

INTERVENTIONS:
Behavioral: Beating the Blues — Automated, cognitive behavioral therapy delivered via a website. There are 8 sessions, each taking one to 1.5 hours to complete. Sessions are prerecorded and sequenced. Sessions are based on the principles of cognitive behavioral therapy and include techniques such as cognitive restructuring and behavioral activation. The entire program takes about 8 to 12 weeks to complete.
  Other Names: Internet based cognitive behavioral therapy

SUMMARY:
Depression is one of the most common and debilitating conditions among older adults. At-home seniors, also called homebound seniors, are older adults who are confined to a bed or chair and are unable to get about outdoors. Internet-based CBT (iCBT) delivers CBT via websites or dedicated apps on mobile devices or tablets. iCBT can be self-administered or guided by a therapist. Its strengths include low-cost, accessibility, and ability to tailor to individual needs while maintaining fidelity. Despite its potential, iCBT trials have rarely included older adults. Those that included older adults showed that they tended to report more technological challenges but they benefited from the intervention as much as younger adults did. As far as we know, studies have not yet tested the feasibility and preliminary effects of iCBT with a diverse group of at-home seniors receiving non-skilled home care. This study explores the feasibility and acceptability of delivering iCBT to a sample of at-home seniors who receive non-skilled home care. Home care workers who care for these seniors are recruited to provide assistance for completing iCBT. We hypothesize that iCBT is an acceptable and feasible intervention for treating depression among at-home seniors.

DETAILED DESCRIPTION:
Depression is one of the most common and debilitating conditions among older adults. At-home seniors, also called homebound seniors, are older adults who are confined to a bed or chair and are unable to get about outdoors. Medical morbidity, disability, cognitive impairment, pain, and social isolation are known risk factors for depression that are prevalent among at-home seniors. Epidemiological and community-based studies have consistently documented a high prevalence of depression among at-home seniors. However, depression treatment is often inaccessible to at-home seniors. The majority of at-home seniors with depression do not receive adequate treatment, with the dominant treatment modality being medication. Successfully treating late-life depression requires a multi-component treatment program beyond medication. Besides, medication non-adherence is common due to concerns of side effects and preferences for other treatment modalities such as counseling. However, office-based psychotherapy is out of reach for at-home seniors who often require assistance for transportation. In addition, older adults prefer home-based treatment and counseling, and consideration of their preference may lead to better treatment outcomes.

Online therapy (iCBT) is an evidence-based approach for treating depression. Cognitive-behavioral therapy (CBT) is the gold standard of psychotherapy for depression in both young and older adults. Internet-based CBT (iCBT) delivers CBT via d websites or dedicated apps on mobile devices or tablets. iCBT can be self-administered or guided by a therapist. Its strengths include low-cost, accessibility, and ability to tailor to individual needs while maintaining fidelity. Meta-analyses have shown that iCBT is equivalent to face-to-face CBT in its effectiveness for treating depression. Emerging evidence suggests that iCBT may actually be more effective for older adults, because they are more likely to adhere to treatment than their younger counterparts. Despite the benefits of iCBT, most older adults do not use iCBT, possibly due to limited opportunities accessing iCBT programs and technological challenges.

This project explores the feasibility of implementing iCBT in non-skilled home care. Home care workers provide personal care and companionship to older adults in need of assistance with daily activities, housekeeping, medication management, and transportation. Home care is provided full-time, part-time, intermittently, or even around the clock to address the recipient's long-term care needs. Home-based care provides a naturalized and accessible setting, and frequent home visits over an extended period offer opportunities for prolonged engagement and symptom monitoring. Research shows that iCBT programs with human support are more effective than self-guided programs. For at-home seniors, home care workers represent an untapped resource of human support and can be trained to provide technical assistance for at-home seniors with limited computer literacy, addressing technological challenges associated with iCBT use. Moreover, home care workers can facilitate the completion of behavioral activation activities (e.g., drive a client to attend a social activity), which is critical in realizing the effectiveness of CBT. In addition, participation in training and intervention may also benefit the home care workers themselves by improving job satisfaction, pride, and retention. However, Studies have not tested iCBT with at-home seniors receiving home care. Protocols for implementing iCBT in home care also do not exist. Issues regarding screening, supervision, and referrals need to be addressed and standardized. In addition, we need to develop strategies to address implementation barriers at the patient, provider, and organization levels to achieve sustained impact.

This pilot feasibility study is a pragmatic trial of iCBT among a sample of diverse at-home seniors receiving non-skilled home care. Guided by the Replicating Effective Programs framework, this study aims to develop materials to package an existing, evidence-based iCBT program called Beating the Blues for testing in a sample of at-home seniors receiving home care. The primary aim of the study is to test whether iCBT is an acceptable treatment modality for at-home seniors with varying levels of technology competency. An exploratory aim is to examine whether it is feasible to train home care workers to assist seniors with iCBT completion. Findings from this pilot study will gather information regarding barriers to implement iCBT in non-skilled home care at the provider- (home care workers) and the patient- (at-home seniors) levels. If the results from this study are promising, subsequent efforts will be devoted to address implementation barriers at the organizational (home care agencies) level.

The study is a single-group open trial. Study materials (measurements, participant workbook) will be piloted tested with 2 subjects, who will not participate in the full trial. The targeted sample size for the full trial is 28. A sample size of 23 provides a power of 0.95 to detect a significant effect size of d=.8 from paired-sample t-test (G*Power, 3.1 version). A proposed sample size of 28 therefore has sufficient power to detect the projected effect size.

Study subjects will be recruited from home-care agencies, meals-on-wheels, and senior apartment buildings in Ann Arbor and surrounding areas.

After being screened and consented, subjects will receive a comprehensive baseline assessment. Subjects have the choice of receiving assistance from their home care worker, assistance from a member of the research team, or work on the iCBT program on their own. If subjects prefer to work on the iCBT program with their home care workers, their workers will also been consented and receive a training. After their workers finish the required training, subjects will then start treatment. Research team will supply a tablet and prepaid data packages to subjects if they don't have access to a working device or internet package. Subjects are told that they have 3 months to use the online program. Subjects will receive a comprehensive post-test assessment once they complete the entire program or at the end of the 3-month period, whichever occurs first. Subjects will also be asked to participate in a short individual interview during post-test. All assessments with subjects will take place at their home. The structured part of the comprehensive baseline and post-test includes three parts: an online self-administered survey, a clinical interview, and Montreal Cognitive Assessment (MoCA) test for cognitive impairment using the MoCA app. In addition to these scheduled assessments, Beating the Blues, the iCBT program used in the study, has built-in assessments (PHQ-9 and GAD-7) at the start of session 1 and the end of session 3, 5, 7, & 8.

Survey data will be recorded and managed using Qualtrics.

Post-treatment analysis will involve an intention-to-treat design where missing data are addressed by carrying forward data previously collected. Primary outcomes include Patient Health Questionnaire (PHQ-9) for depressive symptoms, number of sessions completed, and program satisfaction/acceptability. Difference in PHQ-9 between session 1 and post-test will be calculated and tested. Session 1 PHQ-9 score will be used to assure consistency in time lapsed up until post-test. Secondary outcomes include Generalized Anxiety Disorder (GAD-7) for anxiety and Montreal Cognitive Assessment (MoCA) for cognitive impairment. Difference in GAD-7 between session 1 and post-test will be calculated and tested. Difference in MoCA score between baseline and post-test will be tested. Paired-sample t-test will be used to detect statistically significant difference. Effect sizes (Cohen's d) and 95% confidence intervals will be calculated. Statistical analyses will be conducted using Stata 15.1 SE version.

This study is supported by an Investigator-Initiated Grant from the Blue Cross Blue Shield of Michigan Foundation and a grant from the Michigan Department of Health and Human Services.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age

  * have received home care for ≥ 1 month and anticipate continued care for ≥ 3 months
  * have at least mild depressive symptoms (PHQ-9≥5)
  * speak English.

Exclusion Criteria:

* Currently receiving psychotherapy
* Have a psychotic disorder (BPRS)
* Have active suicidal ideation based on endorsement of PHQ-9 item 9 (other than not at all)
* Severe cognitive impairment, assessed as having ≥ 3 errors on the 6-item Mini mental state exam
* Have a planned hospital admission in the next 3 months of enrollment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 Items (PHQ-9) | Change from baseline PHQ9 at end of treatment (3 months after the start of treatment)
  PHQ-9 for depressive symptoms, total score ranges from 0 to 27, higher scores indicate worse depressive symptoms
# of sessions completed | Up to 3 months after the start the treatment
  # of Beating the Blues sessions completed at the end of 3 months
Acceptability | Up to 3 months after the start the treatment
  Treatment acceptability scale, has a total of 10 questions, total score ranges from 10 to 50, higher scores indicate higher acceptability
Satisfaction with the treatment program | Up to 3 months after the start the treatment
  self rated satisfaction with the program, score ranges from 1 to 10. Higher score indicates higher satisfaction.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | Change from baseline GAD7 at end of treatment (3 months after the start of treatment)
  Anxiety symptoms assessment, total score ranges from 0 to 21, higher score indicating worse anxiety symptoms
Montreal Cognitive Assessment (MoCA) | Change from baseline MoCA at end of treatment (3 months after the start of treatment)
  Cognitive impairment assessment. Total score ranges from 0 to 30. Higher score indicates better cognition and less cognitive impairment.
EQ5D-5L | Change from baseline EQ5D at end of treatment (3 months after the start of treatment)
  This measures health related quality of life. EQ5D-5L has five questions and total score is not a simple sum of questions. Scores needs to be converted into utility scores based on population norms. Final utility index score ranges from 0 to 1 (1-sum of raw utility scores), with a higher score indicating better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoling Xiang, PhD, MSW, Principal Investigator — University of Michigan School of Social Work
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiang X, Kayser J, Sun Y, Himle J. Internet-Based Psychotherapy Intervention for Depression Among Older Adults Receiving Home Care: Qualitative Study of Participants' Experiences. JMIR Aging. 2021 Nov 22;4(4):e27630. doi: 10.2196/27630. PMID 34813491